CLINICAL TRIAL: NCT02883517
Title: Detection of Somatic Mutations on Cell-free Circulating DNA in Potentially Aggressive Cutaneous Lymphomas
Brief Title: Cell-free Circulating DNA in Primary Cutaneous Lymphomas
Acronym: MATULILA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2015/35
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Mycosis Fungoides; Lymphoma, Large B-cell, Diffuse
Keywords: cell-free circulating DNA;; digital PCR; liquid biopsy
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a collection of plasma collected at different times during the management of patients with aggressive cutaneous lymphomas followed at the University Hospital of Bordeaux.
  Collection of tumor tissue biopsies for Next Generation Sequencing analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aggressive primary cutaneous lymphomas: * Mycosis fungoides ≥ T2b
  * Primary cutaneous T helper follicular lymphoma ≥ T2
  * Primary cutaneous diffuse large B-cell lymphoma, leg type Genetic: Cytogenetic and molecular studies Detect cell-free circulating tumoral DNA in a blood sample, with correlations with clinical characteristics and metastatic outcome.
  Interventions: Genetic: Cytogenetic and molecular studies

INTERVENTIONS:
Genetic: Cytogenetic and molecular studies — Detect cell-free circulating tumoral DNA in a blood sample, with correlations with clinical characteristics and metastatic outcome.

SUMMARY:
To evaluate the possibility of detecting cell-free circulating tumoral DNA in potentially aggressive primary cutaneous lymphomas, the investigator opted to search a representative tumor sample mutation in the blood of these patients, by digital PCR. Patients with mycosis fungoides, primary cutaneous T-cell lymphoma helper follicular phenotype and primary cutaneous diffuse large B-cell lymphoma, leg-type will be included and 4 blood samples will be collected during 12 months.

DETAILED DESCRIPTION:
Primary cutaneous lymphomas represent the second extra nodal localization of lymphomas, and are constituted by T-cell and B-cell phenotype lymphomas. Mycosis fungoides, a T-cell epidermotropic lymphoma, is the most frequent. Its clinical behavior is usually indolent but some patients have an aggressive evolution. Among B-cell cutaneous lymphomas, primary cutaneous diffuse large B-cell lymphoma, leg type (PCDLBCL-LT) is the most aggressive. Cytogenetic and molecular studies on these tumours led to a genetic characterization of these entities. Therefore, there is not any biologic marker that can help monitoring these lymphomas. In solid tumors, mutations exhibited by the tumour tissue has been detected in plasma of patients, assessing the possibility to detect cell-free circulating tumoral DNA in a blood sample, with correlations with clinical characteristics and metastatic outcome. The concept of liquid biopsies, allowing the detection of tumour mutation in plasma has been validated in nodal diffuse large B-cell lymphoma. That's why the purpose is to evaluate the possibility to detect cell-free circulating tumoral DNA in primary cutaneous lymphomas, using a highly sensitive method (digital PCR), combined with a next generation sequencing panel of the tumour sample.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* French social security system affiliation or equivalent;
* Patient with an aggressive cutaneous lymphoma (PCDLBCL-LT, mycosis fungoides, T helper follicular cutaneous lymphoma) diagnosed and monitored at the university hospital of Bordeaux;
* Written and informed consent obtained for genetic blood test;
* Biopsy sample available for molecular analysis.

Exclusion Criteria:

* Another cancer (except "in situ" and surgery treated cutaneous carcinomas) in the precedent 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an aggressive cutaneous Lymphomas
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have circulating free tumor DNA (detected by Digital polymerase chain reaction) with the mutation identified on biopsy | Day 1
Proportion of patients who have circulating free tumor DNA (detected by Digital polymerase chain reaction) with the mutation identified on biopsy | Week 12
Proportion of patients who have circulating free tumor DNA (detected by Digital polymerase chain reaction) with the mutation identified on biopsy | Week 24
Proportion of patients who have circulating free tumor DNA (detected by Digital polymerase chain reaction) with the mutation identified on biopsy | Week 36

SECONDARY OUTCOMES:
Amount of circulating tumor DNA (number of copies / µl) | Day 1
Amount of free circulating DNA (number of copies / µl) | Day 1
Number of patient with presence or absence of blood lymphocyte clone identical to the tumor clone | Day 1
Number of patient with presence or absence of blood lymphocyte clone identical to the tumor clone | Week 12
Number of patient with presence or absence of blood lymphocyte clone identical to the tumor clone | Week 24
Number of patient with presence or absence of blood lymphocyte clone identical to the tumor clone | Week 36
Number of patient with presence or absence of mutation identified in circulating blood | Day 1
Number of patient with presence or absence of mutation identified in circulating blood | Week 12
Number of patient with presence or absence of mutation identified in circulating blood | Week 24
Number of patient with presence or absence of mutation identified in circulating blood | Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Anne PHAM-LEDARD, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux - Hospital Saint André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No